CLINICAL TRIAL: NCT03828734
Title: Modulation of Alpha and Theta Oscillations in a Cognitive Control Retrospective Cue Task With Frequency Specific Rhythmic Transcranial Magnetic Stimulation
Brief Title: Modulation of Cognitive Control Signals in Prefrontal Cortex by Rhythmic Transcranial Magnetic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18-1789; R01MH111889 (NIH)
Record Dates: First submitted 2019-01-29; First posted 2019-02-04 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2019-12

CONDITIONS: Executive Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TMS to frontal cortex followed by TMS to parietal cortex (Experimental): Participants will receive TMS while performing a cognitive control task. In their first stimulation session, the TMS coil will be placed over the frontal cortex on the scalp. In their second session, the TMS coil will be placed over the parietal cortex on the scalp. During every session, subjects receive Theta TMS, Alpha TMS, and Arrhythmic TMS.
  Interventions: Device: Theta TMS; Device: Alpha TMS; Device: Arrhythmic TMS
- TMS to parietal cortex followed by TMS to frontal cortex (Experimental): Participants will receive TMS while performing a cognitive control task. In their first stimulation session, the TMS coil will be placed over the parietal cortex on the scalp. In their second session, the TMS coil will be placed over the frontal cortex on the scalp. During every session, subjects receive Theta TMS, Alpha TMS, and Arrhythmic TMS.
  Interventions: Device: Theta TMS; Device: Alpha TMS; Device: Arrhythmic TMS

INTERVENTIONS:
Device: Theta TMS — TMS will be administered at the frequency of each subject's endogenous theta oscillation (4-7Hz)
  Other Names: MagProX100
Device: Alpha TMS — TMS will be administered at the frequency of each subject's endogenous alpha oscillation (8-12 Hz)
  Other Names: MagProX100
Device: Arrhythmic TMS — TMS will be administered arrhythmically; i.e. a sequence of pulses with randomized timing
  Other Names: MagProX100

SUMMARY:
Purpose: In this study, the investigators will provide causal evidence for the role of alpha and theta oscillations in cognitive control.

Participants: Participants must be healthy, between the ages of 18 and 35, right handed, able to provide informed consent, willing to comply with all study procedures, and be available for the duration of the study, speak and understand English.

Procedures: Alpha and theta brain oscillations will be measured and then entrained using frequency specific rhythmic TMS during a retrospective cued cognitive control task.

DETAILED DESCRIPTION:
Neural oscillations are proposed to be a mechanism of coordinating information processing across distributed regions of cortex. Different neural oscillations may correspond to different underlying neural computations. Noninvasive brain stimulation allows experimenters to modulate specific neural oscillations by targeting particular frequency bands. By collecting simultaneous electroencephalography (EEG), rhythmic transcranial magnetic stimulation (TMS) has been previously demonstrated to entrain neural oscillations at the frequency of stimulation. Furthermore, when the frequency of entrained neural oscillations is matched to the frequency of endogenous activity in a cognitive task, the brain stimulation improves behavioral performance. Therefore, noninvasive brain stimulation is a promising tool for improving cognition by inducing optimal neural activity via externally applied electromagnetic fields; e.g. cognitive control improvements.

Previous evidence has implicated neural activity in the alpha band (8-12 Hz) in information suppression and activity in the theta band (4-7 Hz) in information prioritization. Cognitive control task paradigms have been shown to elicit distinct activity in both of these bands. In this task, the stimuli are lateralized to the right and left visual field during encoding. After a short delay, a cue informs participants which stimuli (right or left) will be tested. Previous evidence found that alpha activity in parietal cortex is generated contralateral to irrelevant stimuli-supporting the role of alpha in information suppression-while theta activity in frontal cortex increases with the number of stimuli to be remembered-supporting the role of theta in information prioritization.

For the current study, the investigators propose to deliver rhythmic trains of TMS in either alpha frequency, theta frequency, or an arrhythmic control to modulate neural processing during a cognitive control task. By collecting simultaneous EEG with TMS, the investigators will be able to measure the entrained oscillations from rhythmic TMS. The goal of this experiment is to enhance the observed theta and alpha activity that is seen with the successful prioritization and suppression of information. To provide causal evidence that parietal cortex generates alpha activity and frontal cortex generates theta activity, the investigators will apply rhythmic TMS stimulation to two scalp locations: the anterior middle frontal gyrus and inferior intraparietal sulcus. By applying alpha frequency, theta frequency, and arrhythmic TMS at each location, the investigators will be able to examine the causal relationship of frontal theta oscillations in information prioritization and parietal alpha oscillations in information suppression.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Between the ages of 18 and 35
* Right handed
* Able to provide informed consent
* Willing to comply with all study procedures
* Available for the duration of the study
* Speak and understand English.

Exclusion Criteria:

* Attention Deficit Hyperactivity Disorder (currently under treatment)
* Neurological disorders and conditions, including, but not limited to: History of epilepsy Seizures (except childhood febrile seizures) -Dementia
* History of stroke
* Parkinson's disease
* Multiple sclerosis
* Cerebral aneurysm
* Brain tumors
* Medical or neurological illness or treatment for a medical disorder that could interfere with study participation (e.g., unstable cardiac disease, HIV/AIDS, malignancy, liver or renal impairment)
* Prior brain surgery -Any brain devices/implants, including cochlear implants and aneurysm clips -Cardiac pacemaker -Any other implanted electronic device -History of current traumatic brain injury -(For females) Pregnancy or breast feeding -Anything that, in the opinion of the investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Albouy P, Weiss A, Baillet S, Zatorre RJ. Selective Entrainment of Theta Oscillations in the Dorsal Stream Causally Enhances Auditory Working Memory Performance. Neuron. 2017 Apr 5;94(1):193-206.e5. doi: 10.1016/j.neuron.2017.03.015. Epub 2017 Mar 23. PMID 28343866
- [Background] Roux F, Uhlhaas PJ. Working memory and neural oscillations: alpha-gamma versus theta-gamma codes for distinct WM information? Trends Cogn Sci. 2014 Jan;18(1):16-25. doi: 10.1016/j.tics.2013.10.010. Epub 2013 Nov 19. PMID 24268290
- [Background] Fries P. Rhythms for Cognition: Communication through Coherence. Neuron. 2015 Oct 7;88(1):220-35. doi: 10.1016/j.neuron.2015.09.034. PMID 26447583
- [Background] Hanslmayr S, Matuschek J, Fellner MC. Entrainment of prefrontal beta oscillations induces an endogenous echo and impairs memory formation. Curr Biol. 2014 Apr 14;24(8):904-9. doi: 10.1016/j.cub.2014.03.007. Epub 2014 Mar 27. PMID 24684933
- [Background] Klimesch W, Sauseng P, Hanslmayr S. EEG alpha oscillations: the inhibition-timing hypothesis. Brain Res Rev. 2007 Jan;53(1):63-88. doi: 10.1016/j.brainresrev.2006.06.003. Epub 2006 Aug 1. PMID 16887192
- [Background] Popov T, Popova P, Harkotte M, Awiszus B, Rockstroh B, Miller GA. Cross-frequency interactions between frontal theta and posterior alpha control mechanisms foster working memory. Neuroimage. 2018 Nov 1;181:728-733. doi: 10.1016/j.neuroimage.2018.07.067. Epub 2018 Jul 31. PMID 30075276
- [Background] Reinhart RMG. Disruption and rescue of interareal theta phase coupling and adaptive behavior. Proc Natl Acad Sci U S A. 2017 Oct 24;114(43):11542-11547. doi: 10.1073/pnas.1710257114. Epub 2017 Oct 9. PMID 29073084
- [Background] Romei V, Thut G, Silvanto J. Information-Based Approaches of Noninvasive Transcranial Brain Stimulation. Trends Neurosci. 2016 Nov;39(11):782-795. doi: 10.1016/j.tins.2016.09.001. Epub 2016 Sep 30. PMID 27697295
- [Background] Thut G, Veniero D, Romei V, Miniussi C, Schyns P, Gross J. Rhythmic TMS causes local entrainment of natural oscillatory signatures. Curr Biol. 2011 Jul 26;21(14):1176-85. doi: 10.1016/j.cub.2011.05.049. Epub 2011 Jun 30. PMID 21723129
- [Background] Wallis G, Stokes M, Cousijn H, Woolrich M, Nobre AC. Frontoparietal and Cingulo-opercular Networks Play Dissociable Roles in Control of Working Memory. J Cogn Neurosci. 2015 Oct;27(10):2019-34. doi: 10.1162/jocn_a_00838. Epub 2015 Jun 4. PMID 26042457
- [Background] Wang XJ. Neurophysiological and computational principles of cortical rhythms in cognition. Physiol Rev. 2010 Jul;90(3):1195-268. doi: 10.1152/physrev.00035.2008. PMID 20664082
- [Background] Wolinski N, Cooper NR, Sauseng P, Romei V. The speed of parietal theta frequency drives visuospatial working memory capacity. PLoS Biol. 2018 Mar 14;16(3):e2005348. doi: 10.1371/journal.pbio.2005348. eCollection 2018 Mar. PMID 29538384
- [Background] Rouder JN, Morey RD, Morey CC, Cowan N. How to measure working memory capacity in the change detection paradigm. Psychon Bull Rev. 2011 Apr;18(2):324-30. doi: 10.3758/s13423-011-0055-3. PMID 21331668

RESULTS

PARTICIPANT FLOW:
Groups:
- TMS to Frontal Cortex Followed by TMS to Parietal Cortex: Participants will receive transcranial magnetic stimulation (TMS) while performing a cognitive control task. In the first stimulation session, the TMS coil will be placed over the frontal cortex on the scalp. In the second session, the TMS coil will be placed over the parietal cortex on the scalp. During every session, participants receive Alpha TMS, Theta TMS, and Arrhythmic TMS.
- TMS to Parietal Cortex Followed by TMS to Frontal Cortex: Participants will receive TMS while performing a cognitive control task. In their first stimulation session, the TMS coil will be placed over the parietal cortex on the scalp. In their second session, the TMS coil will be placed over the frontal cortex on the scalp. During every session, participants receive Alpha TMS, Theta TMS, and Arrhythmic TMS.
Period: Baseline
Arm/Group | TMS to Frontal Cortex Followed by TMS to Parietal Cortex | TMS to Parietal Cortex Followed by TMS to Frontal Cortex
Started | 32 | 26
Completed | 32 | 26
Not Completed | 0 | 0
Period: Pre-Randomization (1 Week)
Arm/Group | TMS to Frontal Cortex Followed by TMS to Parietal Cortex | TMS to Parietal Cortex Followed by TMS to Frontal Cortex
Started | 32 | 26
Completed | 29 | 25
Not Completed | 3 | 1
Period: First Intervention
Arm/Group | TMS to Frontal Cortex Followed by TMS to Parietal Cortex | TMS to Parietal Cortex Followed by TMS to Frontal Cortex
Started | 29 | 25
Completed | 25 | 25
Not Completed | 4 | 0
Period: First Washout (1 Week)
Arm/Group | TMS to Frontal Cortex Followed by TMS to Parietal Cortex | TMS to Parietal Cortex Followed by TMS to Frontal Cortex
Started | 25 | 25
Completed | 25 | 24
Not Completed | 0 | 1
Period: Second Intervention
Arm/Group | TMS to Frontal Cortex Followed by TMS to Parietal Cortex | TMS to Parietal Cortex Followed by TMS to Frontal Cortex
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants will receive TMS while performing a cognitive control task. In one stimulation session, the TMS coil will be placed over the frontal cortex on the scalp. In another session, the TMS coil will be placed over the parietal cortex on the scalp. During every session, participants receive Alpha TMS, Theta TMS, and Arrhythmic TMS.
Arm/Group | All Participants
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.2 (3.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 31
  More than one race | 3
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 58
Number of Remembered Items [Mean (Standard Deviation); unit: number of remembered items] — Participants make a button press on a keyboard to indicate if the probed items are matched or non-matched to the items held in memory after a retrospective cue. The percent correct for non-match conditions is defined as the hit rate, and the percent incorrect for match condition is defined as the false alarm rate. The number of remembered items, often referred to as working memory capacity, is calculated as the number of items presented (2, 3, or 4) times the hit rate minus the false alarm rate, divided by one minus false alarm rate. Range of values is 0 to 4 where larger is better.
  number of remembered items | 1.8039 (0.4988)
Response Time [Mean (Standard Deviation); unit: seconds] — Participants make a button press on a keyboard to indicate if the probe items are matched or non-matched to the items held in memory after a retrospective cue is presented. The investigators will calculate the response time of this choice as the difference between the time of the button press and presentation of the probe. A faster response time represents better performance.
  seconds | 0.8225 (0.1605)

OUTCOME MEASURES:

1. Primary Outcome: Number of Remembered Items
Description: Participants make a button press on a keyboard to indicate if the probed items are matched or non-matched to the items held in memory after a retrospective cue is presented. The investigators calculate the percent correct for non-match conditions, defined as the hit rate, and the percent incorrect for match conditions, defined as the false alarm rate. The number of remembered items, often referred to as working memory capacity, is calculated as the number of items to be remembered (2, 3, or 4) times the hit rate minus the false alarm rate, divided by one minus the false alarm rate. The range of values is 0 to 4 where larger values mean better performance. For TMS to frontal cortex, working memory capacity is reported when the participant was cued to the right. For TMS to parietal cortex, working memory capacity is reported when the participant was cued to the left.
Time Frame: 1 week
Population: 54 participants were randomized into the experiment arms. 5 participants did not complete both arms and are excluded from analysis. In addition, data from 2 participant was corrupted and 5 participants were excluded due to poor task performance. Analysis was run on 42 participants.
Measure: Mean (Standard Deviation); unit: number of remembered items
Groups:
- TMS to Frontal Cortex: Participants receive TMS to frontal cortex while performing a cognitive control task. During every session, participants receive Theta TMS, Alpha TMS, and Arrhythmic TMS.
- TMS to Parietal Cortex: Participants receive TMS to parietal cortex while performing a cognitive control task. During every session, participants receive Theta TMS, Alpha TMS, and Arrhythmic TMS.
Arm/Group | TMS to Frontal Cortex | TMS to Parietal Cortex
Number analyzed (Participants) | 42 | 42
number of remembered items
  Theta TMS | 1.863 (0.613) | 1.754 (0.524)
  Alpha TMS | 1.796 (0.495) | 1.797 (0.572)
  Arrhythmic TMS | 1.803 (0.381) | 1.864 (0.469)
Statistical Analysis 1: Comparison: TMS to Frontal Cortex vs TMS to Parietal Cortex; Test type: Superiority; p = 0.263, ANOVA

2. Primary Outcome: Amplitude of Neural Oscillations
Description: The electrical activity of the brain is recorded during performance of the task and brain stimulation. The investigators will perform Morlet wavelet convolution on the recorded electrical signal to calculate the amplitude of neural oscillations in the frequency bands: theta (4-7 hertz) and alpha (8-12 hertz). The amplitude of neural oscillations is reported during the second half of stimulation in the region that is being stimulated. The amplitude is normalized for each participant as the percent change from the amplitude during the baseline period (before the task begins). For TMS to frontal cortex the amplitude of theta oscillations are reported and for TMS to parietal cortex the amplitude of alpha oscillations are reported.
Time Frame: 1 week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | TMS to Frontal Cortex | TMS to Parietal Cortex
Number analyzed (Participants) | 42 | 42
microvolts
  Theta TMS | 1.443 (1.227) | -0.201 (0.505)
  Alpha TMS | 0.489 (0.412) | 0.241 (1.045)
  Arrhythmic TMS | 0.944 (0.705) | -0.132 (0.600)
Statistical Analysis 1: Comparison: TMS to Frontal Cortex vs TMS to Parietal Cortex; Test type: Superiority; p < 0.000001, ANOVA

3. Primary Outcome: Response Time
Description: Participants make a button press on a keyboard to indicate if the probe items are matched or non-matched to the items held in memory after a retrospective cue is presented. The investigators will calculate the response time of this choice as the difference between the time of the button press and presentation of the probe. For TMS to frontal cortex, response time is reported when the participant was cued to the right. For TMS to parietal cortex, response time is reported when the participant was cued to the left.
Time Frame: 1 week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | TMS to Frontal Cortex | TMS to Parietal Cortex
Number analyzed (Participants) | 42 | 42
seconds
  Theta TMS | 0.728 (0.157) | 0.714 (0.154)
  Alpha TMS | 0.711 (0.162) | 0.710 (0.162)
  Arrhythmic TMS | 0.720 (0.155) | 0.717 (0.166)
Statistical Analysis 1: Comparison: TMS to Frontal Cortex vs TMS to Parietal Cortex; Test type: Superiority; p = 0.399, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were systematically assessed after the 3 hour session for both arms. Each session was 1 week apart. Thus, adverse events were monitored for approximately 1 week.
Arm/Group | TMS to Frontal Cortex | TMS to Parietal Cortex
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/50
Other Adverse Events (participants affected / at risk) | 25/53 | 25/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMS to Frontal Cortex (N=53) | TMS to Parietal Cortex (N=50)
Headache (Skin and subcutaneous tissue disorders) | 11 (11) | 11 (11)
Neck pain (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 9 (9) | 8 (8)
Tingling (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Ringing or buzzing noise (Ear and labyrinth disorders) | 0 (0) | 0 (0)
Burning sensation (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Local redness (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Sleepiness (General disorders) | 10 (10) | 9 (9)
Trouble concentrating (General disorders) | 11 (11) | 6 (6)
Dizziness (General disorders) | 2 (2) | 0 (0)
Flickering lights (General disorders) | 0 (0) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT03828734/Prot_SAP_000.pdf